CLINICAL TRIAL: NCT05781165
Title: Application of Augmented Reality (AR) in HIV Self-test in Men Who Have Sex With Men Community
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tsz Ho Kwan, Research Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: MSS346R
Record Dates: First submitted 2023-03-01; First posted 2023-03-23 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention arm will be able to access the augmented reality page in the web app to perform the HIV self-test
  Interventions: Other: Augmented reality
- Control (No Intervention): Participants in the control arm will be asked to follow the instruction sheet to perform the HIV self-test

INTERVENTIONS:
Other: Augmented reality — Step-by-step 3D models displayed with augmented reality guiding the self-test procedures
  Arms: Intervention

SUMMARY:
Objective: To apply augmented reality (AR) technology in HIV self-test and to assess its impacts in enhancing testing performance among men who have sex with men (MSM).

Design: Parallel randomised controlled, open label, trial. Block randomisation with a block size of 4 would be used to allocate the study arms.

Participants: men who have sex with men in Hong Kong

Intervention: Self-test assisted by AR vs self-test with instruction sheets

Main outcome measures: Effectiveness, usability, learnability, efficiency and satisfaction scores; rate of completion and result upload; acceptability of AR approach in assisting self-test

Anticipated results: 200 MSM would be recruited with 50 and 150 in control and intervention group, respectively. The scores in the intervention group are 10% higher than the control group. Proportion of satisfied participants in the intervention group is 10% more than the control group. AR approach is feasible and acceptable to MSM for assisting in HIV self-test.

DETAILED DESCRIPTION:
About 200 MSM would be recruited through community-based organisations and Internet channels where MSM socialise and seek partners. Fifty and 150 participants would be randomly assigned into the control and intervention group by block randomisation with a block size of 4, respectively. After giving informed consent, subjects would be invited to complete an online questionnaire and request for an HIV self-test kit in the online portal before randomisation. Participants in the control group would be given a standard commercially available self-test kit which included bilingual instruction sheets. Subjects in the intervention arm would be asked to use the AR element to assist the same standard commercially available self-test kit. All participants would be asked to upload the test result and complete a post-test questionnaire on the usability of the test and the AR approach. The result would be validated by an experienced research staff. Subjects with a positive result would be contacted for follow up. Main outcome measures in this study would include the confidence in performing the self-test and the usability of HIV self-testing between the two arms.

ELIGIBILITY:
Inclusion Criteria:

* Adult men who have sex with men
* Has access to a smartphone with internet access

Exclusion Criteria:

* Unable to communicate in written Chinese or English
* Unable to give informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Confidence in performing the self-test | Month 3
  Confidence in performing the self-test in a Likert scale of 1 (least confident) to 10 (most confident)

SECONDARY OUTCOMES:
Usability of the augmented reality web app | Month 3
  Score measured by system usability scale ranged from 0 to 100 (higher scores mean more usable)
Usability of the augmented reality web app | Month 3
  Score measured by single ease question ranged from 1 to 7 (higher scores mean easier)
Usability of the augmented reality web app | Month 3
  Score measured by after scenario questionnaire (average score of the 3-item questionnaire ranged from 1 to 7, higher scores mean more usable)
Usability of the augmented reality web app | Month 3
  Score measured by subjective mental effort questionnaire ranged from 0 to 150 (higher scores mean more difficult)

CONTACTS AND LOCATIONS:
Overall Officials: Tsz Ho Kwan, PhD, Principal Investigator — Jockey Club School of Public Health and Primary Care